## Antidepressant Response in Older Adults with Comorbid PTSD and MDD

Protocol ID 8111 NCT04697693

Statistical Analysis Plan

Document Version Date: January 29th, 2021

## Statistical Analysis

Descriptive statistics for the sample at baseline will be computed and reported in terms of means with standard deviations. The hypotheses under investigation are that (1) individuals with comorbid PTSD and MDD will experience significant depressive symptom improvement with antidepressant treatment and that (2) cognitive and physical functioning will likewise significantly improve following antidepressant treatment. To investigate these hypotheses, paired samples t-tests will be used to analyze the within-subject change from pre- to post-treatment on depressive symptom severity (Hamilton Rating Scale for Depression [HRSD]), cognitive functioning (NIH Toolbox total score), and physical functioning (gait speed).